CLINICAL TRIAL: NCT02877563
Title: Contrast Ultrasound Assessment of Perfusion Changes After Peripheral Artery Revascularization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Other Study IDs: 16395
Record Dates: First submitted 2016-08-20; First posted 2016-08-24 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; contrast enhanced ultrasound
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PAD: Patients with PAD who are to undergo surgical or percutaneous revascularization.
  Interventions: Other: Contrast ultrasound perfusion imaging of the limb

INTERVENTIONS:
Other: Contrast ultrasound perfusion imaging of the limb — Contrast enhanced ultrasound imaging at rest and during contractile exercise will be performed prior to revascularization and 3-4 weeks after revascularization.

SUMMARY:
This study represents an important step to validate the use of contrast-enhanced ultrasound (CEU) as a clinical research tool that can be used as a biologic readout of new therapies for Peripheral Artery Disease (PAD), and as a clinically-reasonable method for assessing impact of revascularization. The primary aim is to establish that CEU limb perfusion imaging can be used to accurately assess therapeutic improvements in tissue perfusion that are linked to symptom improvement.

DETAILED DESCRIPTION:
The study will be performed in patients with known history of PAD that are scheduled to undergo either surgical or percutaneous revascularization. Limb rest-stress CEU perfusion imaging will be performed before and 3-4 weeks after revascularization. Quantitative measurements of pre-revascularization perfusion, post-revascularization perfusion, and change in perfusion will be compared to symptom status (Rutherford classification and PAD [Criqui] questionnaire) at each study point, and to data on time to onset of claudication on an upright treadmill exercise study (Gardiner protocol). Results of angiography will be scored and allow determination of the relationship between angiographic severity of disease and exercise perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. History of symptomatic PAD
2. Rutherford score <6
3. Age ≥18 y.o.
4. Scheduled to undergo surgical or percutaneous revascularization

Exclusion Criteria:

1. Major medical illness affecting the limb other than PAD (muscle disease, neuromuscular disease, blood diseases).
2. Pregnant or lactating females (- HCG in women of child bearing age)
3. Hypersensitivity to any ultrasound contrast agent
4. Evidence right-to-left, bi-directional, or transient cardiac shunt; unexplained pulmonary hypertension (PA systolic pressure >40 mm Hg) or more than moderate reduction in left ventricular systolic function identified on screening echo.
5. Allergy to eggs
6. Inability to perform modest plantar flexion exercise

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atherosclerotic peripheral artery disease scheduled to undergo surgical or percutaneous revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle perfusion during exercise stress | 1 month
  Calf skeletal muscle perfusion will be assessed by contrast-enhanced ultrasound during calf raise exercise (every 3 seconds for 30 seconds). This assessment will be performed before and 3-4 weeks after revascularization.

SECONDARY OUTCOMES:
Skeletal muscle perfusion at rest. | 1 month
  Calf skeletal muscle perfusion will be assessed by contrast-enhanced ultrasound at rest. This assessment will be performed before and 3-4 weeks after revascularization.

OTHER OUTCOMES:
Time to claudication on treadmill exercise test | 1 month
  Time to development of claudication for each leg will be determined on an upright treadmill walking exercise study

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No